CLINICAL TRIAL: NCT06538545
Title: The Effect Of Sitting Position On The Labor Process
Acronym: POSİTİON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Hilal Guveri, Principal Investigator, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-04/01
Record Dates: First submitted 2024-07-24; First posted 2024-08-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Bleeding; Pain
Keywords: Bleeding; pregnant; labor duration; pain; Sitting Position
MeSH Terms: conditions — Hemorrhage; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1:Vertical Position (Experimental Group-Primiparous) (Experimental): All pregnant women in the experimental group were allowed to use a sitting position (sitting and rocking on a pilates ball or sitting on a bed) from the active phase until labor. They were allowed to lie down for 10-15 minutes when they were tired or when monitoring or intervention was needed.
  Interventions: Behavioral: Sitting position is used in Experimental Arms 1-2
- Arm 2: Vertical Position (Experimental Group-Multiparous) (Experimental): All pregnant women in the experimental group were allowed to use a sitting position (sitting and rocking on a pilates ball or sitting on a bed) from the active phase until labor. They were allowed to lie down for 10-15 minutes when they were tired or when monitoring or intervention was needed.
  Interventions: Behavioral: Sitting position is used in Experimental Arms 1-2
- Arm 3: Lithotomy Position (Control Group-Primiparous) (Active Comparator): All pregnant women in the control group were followed up with hospital procedures during labor. From the latent phase until labor, the pregnant woman was followed up with hospital procedures. At the end of the latent and active phases, pain assessment was requested and VAS (Appendix 6) was applied. The 2nd and 3rd stages of labor were performed on a normal delivery table in the lithotomy position.
  Interventions: Behavioral: Sitting position is used in Experimental Arms 1-2
- Arm 4: Lithotomy Position (Control Group-multiparous) (Active Comparator): The hospital procedure was applied to determine the birth rates of all pregnant women in the control group. From the latent stage until the birth, the pregnant woman is followed up by applying the hospital procedure. At the end of the latent and active phases, the alarm results were requested to be evaluated and VAS (Appendix 6) was developed. The 2nd and 3rd stages of labor were performed in the lithotomy positions on the normal delivery table.
  Interventions: Behavioral: Sitting position is used in Experimental Arms 1-2

INTERVENTIONS:
Behavioral: Sitting position is used in Experimental Arms 1-2 — sitting position Comparison of sitting position and lithotomy position in labor
  Other Names: Lithotomy position is used in those with Active Comparison Arm 3-4.

SUMMARY:
This study was conducted to determine the effect of sitting position on the labor process. The randomized controlled experimental study was conducted in the delivery room of Sivas Numune Hospital.

ELIGIBILITY:
1. Inclusion Criteria:

   * Age range: 19-35
   * 38-42 weeks of pregnancy
   * No health problems that would prevent the use of sitting position
   * -Amniotic membranes not ruptured
   * Having a singleton pregnancy
   * Fetus in vertex position
   * Labor occurs with normal spontaneous vaginal delivery
   * No diagnosed chronic physical disease
   * No diagnosed psychiatric disease
   * No risky pregnancy, risky delivery and newborn/fetus
   * No communication problems
   * Voluntarily participating in the research
2. Exclusion Criteria:

   * Only women who gave birth at Sivas Sample Hospital were included in the study
   * Women who gave birth more than two times were not included in the study

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 160 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Visual analog scale is applied starting from the 1st stage of labor and until the end of the 2nd stage.If the VAS value is 10, it means there is a lot of pain, and if it is 0, it means there is no pain. | 1 years
  The effect of sitting positions of pregnant women in the 38-42nd weeks of pregnancy on the birth process

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Hilal Güveri, Sivas, Sivas Merkez
  - Cumhuriyet Üniversitesi, Sivas

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
Time Frame: 1 years